CLINICAL TRIAL: NCT06928376
Title: A Multicenter, Prospective, Randomized Controlled Study of the Standard "3+7" Regimen Versus Venetoclax Combined With CACAG Regimen in Newly Diagnosed Adult Patients With Intermediate- and High-risk Acute Myeloid Leukemia
Brief Title: A Multicenter RCT of "3+7" vs Venetoclax + CACAG in Newly Diagnosed Mid/High-Risk AML Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: First Affiliated Hospital of Harbin Medical University (Other); Yantai Yuhuangding Hospital (Other); Chinese People's Liberation Army Air Force General Hospital (Unknown); The General Hospital of Western Theater Command (Other); 940 Hospital of the People's Liberation Army Joint Logistic Support Force (Other); The 960th Hospital of Joint Logistics Support Force of Chinese People's Liberation Army (Unknown); the First People's Hospital of Jining (Unknown)
Responsible Party: Principal Investigator, Daihong Liu, Director of the Department of Hematology, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2024-3-40-2
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia; First Line Therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Venetoclax Combined With CACAG Regimen (Experimental): The CACAG+Venetoclax regimen has a total treatment period of 1 week, with a treatment cycle every 4 weeks, and a total of 1 course of treatment.
  Chidamide: 30 mg, twice a week, for a total of 2 administrations; Azacitidine: 75 mg/m^2 from day 1 to day 7; Cytarabine (Ara-C): 75-100 mg/m^2 every 12 hours from day 1 to day 7; Aclarubicin: 20 mg/m^2 on days 1, 3, and 5; Recombinant human granulocyte colony-stimulating factor (G-CSF): 300 μg/day, continued until neutrophil recovery and white blood cell count is ≥20,000/μL; Venetoclax: 100 mg on day 1, 200 mg on day 2, 400 mg from day 3 to day 14, when used in combination with azole drugs, the dosage is reduced to 100 mg/day.
  Interventions: Drug: Azacytidine;Cytarabine;Aclacinomycin;Chidamide;Venetoclax;Granulocyte colony-stimulating factor
- "3+7" Regimen (Active Comparator): Idarubicin+cytarabine(IA) regimen or daunorubicin+cytarabine(DA) regimen for newly diagnosed AML.Recipients were randomized and those entering this group received IA or DA induction chemotherapy. With the IA regimen,recipients received idarubicin(8-10 mg/m2) for three days and cytarabine(75-100 mg/m2, every 12 hrs) for seven days. With the DA regimen,recipients received daunorubicin(60 mg/m2)for three days and cytarabine(75-100 mg/m2,every 12 hrs)for seven days.
  Interventions: Drug: "3+7"

INTERVENTIONS:
Drug: Azacytidine;Cytarabine;Aclacinomycin;Chidamide;Venetoclax;Granulocyte colony-stimulating factor — Azacytidine (75 mg/m2/day, days 1 to 7). Cytarabine (75-100 mg/m2 bid, days 1 to 5). Aclacinomycin(20 mg/day, days 1,3,5). Chidamide (30 mg/day , days 1,4,8,11). Venetoclax (400 mg/day, days 1 to 14,Combined with posaconazole reduced to 100 mg/day,Combined with voriconazole reduced to 200 mg/day ).
  Granulocyte colony-stimulating factor (300 μg/day, day 0 until agranulocytosis recovery)
  Other Names: CACAG+VEN
  Arms: Venetoclax Combined With CACAG Regimen
Drug: "3+7" — IA regimen:
  Idarubicin (8-10 mg/m2) for 3 days . Cytarabine (75-100mg/m2, every 12 hrs) for 7 days.
  DA regimen:
  Daunorubicin(60 mg/m2) for 3 days. Cytarabine (75-100mg/m2, every 12 hrs) for 7 days.
  Other Names: IA or DA
  Arms: "3+7" Regimen

SUMMARY:
The purpose of this study is to compare the efficacy and safety of venetoclax combined with the CACAG regimen with the traditional "3+7" regimen in the treatment of newly diagnosed intermediate- or high-risk acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
Despite the availability of hematopoietic stem cell transplantation and the emergence of many new therapeutic drugs, the prognosis of newly diagnosed acute myeloid leukemia is still poor.Over the past years, combination chemotherapy with anthracycline and standard dose cytarabine (standard "3+7" induction therapy) remains the standard induction. In order to improve the outcome of patients with de novo AML, we developed a venetoclax combined with CACAG regimen in the treatment of de novo AML. In this study, we intent to compare the efficacy and safety of venetoclax combined with CACAG regimen with the traditional "3+7" regimen in the treatment of newly diagnosed intermediate- or high-risk acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

Age 14 to 75 years (no gender limitation) Newly diagnosed with intermediate- or high-risk AML (excluding M3) Liver function: ALT and AST ≤ 2.5 times upper limit of normal; bilirubin ≤ 2 times upper limit of normal Renal function: creatinine ≤ upper limit of normal No uncontrolled infections, organ dysfunction, or severe mental illness ECOG performance status score of 0-2 and predicted survival ≥ 4 months No severe allergic constitution

Exclusion Criteria:

Allergy or contraindication to the study drug Pregnant or breastfeeding female patients Known history of alcohol or drug addiction (due to potential non-compliance) Mental illness or conditions preventing protocol compliance Less than 6 weeks after major organ surgery Liver function: ALT and AST > 2.5 times upper limit of normal; bilirubin > 2 times upper limit of normal Renal function: creatinine > upper limit of normal Deemed unsuitable for the clinical trial (poor compliance, substance abuse, etc.)

-

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-04-18 (Estimated); Study Completion 2026-10-18 (Estimated)

PRIMARY OUTCOMES:
Composite Complete Remission (CRc) Rate after 1 course of treatment | 1 months after study treatment
  a combination of complete remission (CR) and complete remission with incomplete blood count recovery (CRi)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) after 1 course of treatment | 1 months after the start of study treatment
  Defined as the percentage of participants achieving a best overall response of complete response (CR), CR with incomplete blood count recovery (CRi), or partial response (PR).Biological characteristics exploratory studies were analyzed by single-cell sequencing and Atac-seq. Further, according to European LeukemiaNet risk group, we analyzed the outcomes of patients by molecular subtype as a sub-group analysis.
Complete Remission (CR) Rate after 1 courses of treatment | after 1 courses of chemotherapy (each course is 28 days)
  Defined in accordance with the IWG Response Criteria in AML. Bone marrow blasts<5 percent; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 109/L (1000/µL); platelet count >100 x 109/L (100,000/µL); independence of red cell transfusions.
Rate of Minimal Residual Disease (MRD)-Negative Response | after each courses of chemotherapy (each course is 28 days)
  Percentage of participants who achieved MRD-negative response, defined as < 1 leukemia cell per 10,000 leukocytes as assessed by flow cytometry.
Event-free survival | 180 days after study treatment
  Defined as the time interval from treatment initiation to the occurrence of induction failure,relapse,or death,whichever came first.
Overall Survival | 180 days after study treatment
  Defined as the time from joining the clinical study to death due to any cause.
Treatment-related adverse events | From the first dose of study treatment to 30 days after the discontinuation of treatment
  Defined as adverse events that occurred from the first dose of study treatment to 30 days after the discontinuation of treatment.
Disease-free survival | 180 days after study treatment
  Defined as the time interval from disease remission to the occurrence of relapse or death,whichever came first.
Early death | Within 30 days of the start of the first course of treatment
  Defined as death within 30 days of chemotherapy.
Complete Remission with Incomplete Blood Count Recovery (CRi)after 1 courses of treatment | after 1 courses of chemotherapy (each course is 28 days)
  Disappearance of leukemia blasts in the bone marrow (<5% blasts) but without full recovery of blood counts (neutrophils <1.0 x 10⁹/L and/or platelets <100 x 10⁹/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
This study plans to share individual participant data (IPD) with qualified researchers after trial completion. The data to be shared include:
  Demographic information: Age, sex, race, etc. Treatment allocation: Assigned treatment group (e.g., venetoclax + CACAG regimen or "3+7" regimen).
  Efficacy data: Primary and secondary endpoint data (e.g., complete remission rate, overall survival).
  Safety data: Adverse events, serious adverse events, etc. Laboratory results: Hematological, biochemical parameters, and other biomarker data.
  Follow-up data: Recurrence status and long-term outcomes during follow-up. Sharing Conditions Data will be shared in a de-identified format to protect participant privacy. Researchers must submit a formal request outlining the purpose and analysis plan.
  Data use is restricted to research purposes only.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This study plans to share individual participant data (IPD) with qualified researchers after trial completion.
Access Criteria: Data will be shared in a de-identified format to protect participant privacy. Researchers must submit a formal request outlining the purpose and analysis plan.
  Data use is restricted to research purposes only.

DOCUMENTS (2):
  • Study Protocol (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT06928376/Prot_000.pdf
  • Informed Consent Form (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/76/NCT06928376/ICF_001.pdf